CLINICAL TRIAL: NCT06465056
Title: Use of Botulinum Toxin A in Direct Eyebrow Lift Scar: a Randomized Controlled Clinical Trial
Brief Title: Use of Botulinum Toxin A in Direct Eyebrow Lift Scar
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Campinas, Brazil (Other); Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Suzana Matayoshi, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 73675523.7.0000.0068
Record Dates: First submitted 2024-05-26; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Skin Scarring; Eyebrow Ptosis
Keywords: Botulinum Toxin A; Direct eyebrow lift; Eyebrow scar
MeSH Terms: conditions — Cicatrix | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Right side treatment (Active Comparator): Patients receive botulinum toxin A in right side eyebrow scar and saline in left side scar.
  Interventions: Drug: Botulinum toxin type A
- Left side treatment (Active Comparator): Patients receive botulinum toxin A in left side eyebrow scar and saline in right side scar.
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin application between 3-14 days after direct eyebrow lift surgery.

SUMMARY:
Prospective, controlled and randomized study in which participants indicated for surgery to direct eyebrow lift will be randomized into two groups. In addition to surgery, the patients will be treated with botulinum toxin in one eyebrow and saline (placebo) in the other site. The patients participate as treatment and placebo at the same time. Assessments will be carried out through non-invasive exams.

DETAILED DESCRIPTION:
A component of eyebrow ptosis, part of the natural aging process, with or without asymmetries, is found in the majority of patients who seek the blepharoplasty procedure.

There are several procedures to address this condition, but none of them is undoubtedly superior to the others. The direct eyebrow lift technique is known for providing good eyebrow suspension, predictable results and relatively low complexity surgery, which can be performed with local anesthesia.

However, the biggest concern for surgeons and patients is the final appearance of the scar, which will be in a visible area of the face. Botulinum toxin A has been used in recent studies precisely to improve the appearance of scars. Previous studies mainly evaluated traumatic lacerations and post-tumor excision reconstructions, obtaining positive results, with an improvement in the appearance of the wounds in patients who used the medication. It is a safe drug, used for several years for other purposes and without serious adverse effects according to these studies.

The objective of this study is to compare the use of botulinum toxin A versus 0.9% saline solution in the healing of direct eyebrow lift surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with indication for direct eyebrow lift surgery.

Exclusion Criteria:

* Vulnerable groups: children, pregnant women and immunosuppressed patients
* Allergy to botulinum toxin A
* Patients under 18 years old
* Women who are breastfeeding
* Patients with muscular/neuromuscular diseases such as myasthenia gravis and amyotrophic lateral sclerosis
* Patients who underwent botulinum toxin A injection in the last 6 months prior to surgery
* Patients with a history of radiotherapy, chemotherapy or hematological disorders
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Scar evaluation 1 | One month, three months and six months after surgery
  Eyebrow direct lift scar evaluation, comparing botulinum toxin A side with saline side, using the following assessment scale: Visual Analogue Scale Score (VAS). The VAS is described as a quick and practical way of evaluating the patient's experience in relation to pain, on a scale of 0 to 100 millimeters, ranging from no pain to the worst pain imaginable.17 Due to the ease and simplicity of its application, it is used in several studies to evaluate various parameters, even if not consistent with their original validation. Here it will be using meaning 0 (no scar) and 100 milimeters (worst scar imaginable).
Scar evaluation 2 | One month, three months and six months after surgery
  Eyebrow direct lift scar evaluation, comparing botulinum toxin A side with saline side, using the following assessment scale: Vancouver Scar Scale (VSS). The VSS ranges from 0 (best) to 13 (worst) points, evaluating vascular distribution, thickness, flexibility and pigmentation.
Scar evaluation 3 | One month, three months and six months after surgery
  Eyebrow direct lift scar evaluation, comparing botulinum toxin A side with saline side, using the following assessment scale: Stony Brook Scar Evaluation Scales (SBSESs). The SBSES was developed for short-term assessment of repaired burns, and is described as useful for assessment of suture scars. It consists of five indicators: length, elevation or depression, color, suture or staple marks and general appearance. Your score ranges from 0 (worst) to 5 (best)
Scar evaluation 4 | One month, three months and six months after surgery
  Eyebrow direct lift scar evaluation, comparing botulinum toxin A side with saline side, using the following assessment scale: Patient and Observer Scar Assessment Scale (POSAS).
  POSAS was developed in 2004 and is the first scale to consider the perspective of the patient and the evaluator. It is useful in evaluating postoperative and linear scars, ranging from 5 (worst) to 50 (best). It encompasses physical properties of scars such as vascularity, pigmentation, thickness, relief and flexibility, in addition to two patient symptoms, pain and itching.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - University of São Paulo (Clinical Hospital), São Paulo
  - Ophthalmology Dept. University of Sao Paulo General Hospital, São Paulo

IPD SHARING:
Plan to Share IPD: No